CLINICAL TRIAL: NCT01492868
Title: My Nose Study: Sinusitis in Children and How Virus Infections Promote Secondary Bacterial Infections
Brief Title: Sinusitis in Children and the Nasopharyngeal Microbiome
Status: Completed | Type: Observational
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Other Study IDs: 2015-0562; 1R01AI097172-01 (NIH); 2011-0535 (Other: HS IRB); GRANT 10785179 (Other: Study Team)
Record Dates: First submitted 2011-12-13; First posted 2011-12-15 (Estimated); Last update posted 2018-05-08 (Actual); Status verified 2018-05

CONDITIONS: Sinusitis
Keywords: sinusitis; upper respiratory infection
MeSH Terms: conditions — Sinusitis; Respiratory Tract Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Nasopharyngeal microbiome samples
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to investigate the relationship between viral infections of the upper respiratory tract, perturbations of the nasopharyngeal microbiome in children, and the risk of acute bacterial sinusitis over a one year period. The investigators will determine the incidence of acute bacterial sinusitis post viral upper respiratory infection and identify the viral antecedent infections and other risk factors which predispose to infection and ultimately design strategies to reduce the burden of disease and antimicrobial resistance.

ELIGIBILITY:
Inclusion Criteria:

* Children 4 to 7 years of age
* Healthy
* English-speaking parent/guardian -

Exclusion Criteria:

* Any underlying condition which would predispose them to the development of sinusitis including congenital or acquired immunodeficiencies
* Craniofacial abnormalities
* Cystic fibrosis
* Allergic rhinitis or a previous episode of chronic sinusitis.

Ages: 4 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Healthy children
Sampling Method: Non-Probability Sample
Enrollment: 323 (Actual)
Dates: Start 2012-01; Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Incidence of acute bacterial sinusitis in children 49 to 84 months of age (which is the peak age incidence of sinusitis) as a complication of an antecedent viral upper respiratory infection. | Over a 1 year time frame

SECONDARY OUTCOMES:
Define relationships between the nasopharyngeal microbiome, viral illnesses, and progression to clinical sinusitis. | Over a 1 year time frame

CONTACTS AND LOCATIONS:
Overall Officials: Ellen R Wald, MD, Principal Investigator — University of Wisconsin, Madison
Locations (2):
- United States (2):
  - UW Pediatrics at 20 S. Park St, Madison, Wisconsin
  - UW Health West Towne Pediatrics, Madison, Wisconsin

REFERENCES:
- See also: University of Wisconsin-Madison Department of Pediatrics Research Information — http://www.pediatrics.wisc.edu/research/

DOCUMENTS (1):
  • Study Protocol (2015-09-03): https://cdn.clinicaltrials.gov/large-docs/68/NCT01492868/Prot_000.pdf